CLINICAL TRIAL: NCT01951508
Title: Effects of Methylphenidate, Modafinil, and MDMA on Emotion-processing in Humans: A Pharmaco-fMRI Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK 36/13
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Healthy; Substance-related Disorder; Mood Disorder
Keywords: Methylphenidate; Modafinil; MDMA; fMRI; emotion-processing; social cognition
MeSH Terms: conditions — Substance-Related Disorders; Mood Disorders | interventions — Methylphenidate; Dexmethylphenidate Hydrochloride; Modafinil; N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylphenidate, Modafinil, MDMA, Placebo (Other): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but four treatment conditions in the same subject.
  Interventions: Drug: Methylphenidate; Drug: Modafinil; Drug: MDMA; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — 60mg per os, single dose
  Other Names: Ritalin; Concerta; Medikinet; Focalin
Drug: Modafinil — 600mg per os, single dose
  Other Names: Modasomil
Drug: MDMA — 125mg per os, single dose
  Other Names: 3,4-Methylenedioxymethamphethamine; Ecstasy
Drug: Placebo — per os
  Other Names: capsules containing manitol looking identical to methylphenidate, modafinil, and MDMA

SUMMARY:
The purpose of this study is to investigate effects of methylphenidate, modafinil, and 3,4-methylenedioxymethamphetamine (MDMA, "Ecstasy") on emotion-processing and cognitive performance using functional magnetic resonance imaging (fMRI) techniques. The primary hypothesis is that these psychostimulants differentially affect processing of emotional stimuli and potentially leading to alterations in social cognition and behavior.

DETAILED DESCRIPTION:
Methylphenidate and modafinil are increasingly used as performance enhancers or "smart drugs" by students. 3,4-methylenedioxymethamphetamine (MDMA, "Ecstasy") is widely used as recreational drug to enhance emotions. We plan to investigate effects of these psychostimulants on emotion-processing and cognitive performance using functional magnetic resonance imaging (fMRI) techniques. Single doses of methylphenidate (60mg), modafinil (600mg), MDMA (125mg), or placebo will be administered before an fMRI scan in a placebo-controlled, randomized cross-over study design in 24 healthy subjects. Subjective emotional effects, sociability, neurohormonal, cardiovascular responses, and plasma drug concentrations will also be assessed and analyzed for potential brain-induced changes in brain activity in networks processing emotions. The primary hypothesis is that these psychostimulants differentially affect processing of emotional stimuli and potentially leading to alterations in social cognition and behavior. The work should clarify the neuropharmacological basis of the potentially differential effects of these drugs. This information will improve our understanding of the neurofunctional effects of methylphenidate, modafinil, and MDMA, and inform the ongoing debate surrounding brain doping with cognitive and mood enhancers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Sufficient understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to refrain from taking illicit psychoactive substances including cannabis during the study
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session, as well as during the study day
* Participants must be willing not to drive a traffic vehicle within 24h following MDMA administration
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session.
* Body mass index: 18-27kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90mmgHg) or Hypotension (SBP<85mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder. This also includes contraindications for MRI scanning (any type of implants such as heart pacer, insulin-pump, cochlea-implants, heart valve)
* Current or previous psychotic or major affective disorder
* Psychotic or major affective disorder in first-degree relatives
* Prior illicit drug use (except tetrahydrocannabinol (THC)-containing products) more than 5 times or any time within the previous 2 months
* Pregnant or nursing women
* Participation in another clinical trial (currently or within the last 30days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc. )
* Tobacco smoking (regularly > 10cigarettes / day)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effect on amygdala and striatum BOLD signal responses to emotional stimuli | 1.5h
  Functional magnetic resonance (MR) images measuring BOLD (blood oxygen level dependency)activity while subjects will be presented with a series of images of human faces, each showing a fearful or a neutral expression, in an event-related design.
Effects on cognitive performance and associated BOLD signal changes in frontal areas | 1.5h
  Functional magnetic resonance (MR) images measuring BOLD (blood oxygen level dependency)activity while subjects perform a response inhibition/attention task.

SECONDARY OUTCOMES:
Subjective effects | 7h
  repeated assessment of subjective effects with validated, standardized questionnaires
Neuroendocrine effects | 7h
  neuroendocrine parameters assessed: prolactin, cortisol, epinephrine, norepinephrine, oxytocin, copeptin
Empathy and social behavior | 7h
  assessment of cognitive and emotional empathy (empathy is going to be assessed by the Multifaceted Empathy Test (MET)), facial emotion recognition (assessed by the Facial Emotion Recognition Task (FERT)), and prosocial behavior (assessed with the Social Value Orientation Test (SVO)).
  , as well as of prosocial behaviour
Physiological effects of methylphenidate, modafinil, and MDMA | 7h
  repeated assessment of blood pressure (mmHg) , heart rate (bpm), body temperature, and pupillary function
Genetic Polymorphisms | 1 day (assessed once after study completion)
  Effects of genetic polymorphisms on the response to methylphenidate, modafinil, and MDMA
Pharmacokinetics of methylphenidate, modafinil, and MDMA | 7h
  Time course of plasma concentration, half-life, pharmacokinetic-pharmacodynamic relationship

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Vizeli P, Liechti ME. Oxytocin receptor gene variations and socio-emotional effects of MDMA: A pooled analysis of controlled studies in healthy subjects. PLoS One. 2018 Jun 18;13(6):e0199384. doi: 10.1371/journal.pone.0199384. eCollection 2018. PMID 29912955
- [Derived] Dolder PC, Muller F, Schmid Y, Borgwardt SJ, Liechti ME. Direct comparison of the acute subjective, emotional, autonomic, and endocrine effects of MDMA, methylphenidate, and modafinil in healthy subjects. Psychopharmacology (Berl). 2018 Feb;235(2):467-479. doi: 10.1007/s00213-017-4650-5. Epub 2017 May 27. PMID 28551715